CLINICAL TRIAL: NCT05963867
Title: An Open-label Phase 1 PET Imaging Trial to Investigate [89Zr]Zr-BI 764532 Biodistribution and Tumour Uptake in Patients With Small-cell Lung Carcinoma or Neuroendocrine Carcinoma
Brief Title: A Study to Test How BI 764532 is Taken up by Tumours in People With Small-cell Lung Cancer or Neuroendocrine Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1438-0004
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Small Cell Lung Carcinoma (SCLC); Neuroendocrine Neoplasms
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental)
  Interventions: Drug: BI 764532; Drug: [89Zr]Zr-BI 764532
- Cohort 2 (Experimental)
  Interventions: Drug: BI 764532; Drug: [89Zr]Zr-BI 764532

INTERVENTIONS:
Drug: BI 764532 — BI 764532
  Other Names: Obrixtamig
Drug: [89Zr]Zr-BI 764532 — [89Zr]Zr-BI 764532

SUMMARY:
This study is open to adults with small cell lung cancer and other neuroendocrine cancers. The study is in people with advanced cancer for whom previous treatment was not successful or no standard treatment exists. The purpose of this study is to find out how a medicine called BI 764532 gets distributed in the body and in tumours.

Participants get BI 764532 when starting treatment. In the first weeks, doctors check how BI 764532 is taken up in tumours by means of an imaging method. If there is benefit for the participants and if they can tolerate it, the treatment is given up to the maximum duration of the study. During this time, participants visit the study site regularly. The total number of visits depends on how they respond to and tolerate the treatment. Doctors record any unwanted effects and regularly check the general health of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Weight ≥ 60kg
* Signed and dated, written informed consent form (ICF) in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to any trial-specific procedures, sampling, or analyses.
* Patient who failed conventional treatment or for whom no therapy of proven efficacy exists or who is not eligible for established treatment options. Patient must have exhausted available treatment options known to prolong survival for their disease. Previous therapies should include at least one line of platinum-based chemotherapy. Previous therapy with anti Programmed Cell Death Protein 1 (PD-1) or Programmed Cell Death Ligand 1 (PD-L1) are allowed.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* At least one evaluable lesion outside of Central Nervous System (CNS) as defined per Response Evaluation Criteria in Solid Tumours (RECIST) 1.1
* Subjects with brain metastases are eligible provided they meet the following criteria:

  * radiotherapy or surgery for brain metastases was completed at least 2 weeks prior to the first administration of BI 764532,
  * patient is off steroids for at least 7 days (physiologic doses of steroids are permitted), and the patient is off anti-epileptic drugs for at least 7 days or on stable doses of anti-epileptic drugs for malignant CNS disease.

Further inclusion criteria apply.

Exclusion Criteria:

* Previous or concomitant malignancies other than the one treated in this trial within the last 2 years except:

  * effectively treated non-melanoma skin cancers
  * effectively treated carcinoma in situ of the cervix
  * effectively treated ductal carcinoma in situ
  * other effectively treated malignancy that is considered cured by local treatment
* Major injuries and/or surgery or bone fracture within 28 days of first dose BI 764532, or planned surgical procedures
* Known leptomeningeal disease or spinal cord compression due to metastatic disease
* Anticoagulant treatment that cannot be safely interrupted based on opinion of the investigator if medically needed
* Active infection that requires medical therapy or other clinically significant intervention
* Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection within 2 weeks prior to study entry (confirmed via polymerase chain reaction (PCR) test or other applicable test as per local requirements) or suspected SARS-CoV-2 infection as per physician assessment, or close contact (within 1 week) with an individual with confirmed SARS-CoV-2 infection
* Any of the following known laboratory evidence of hepatitis virus infection:

  * Positive results of hepatitis B surface (HBs) antigen
  * Presence of hepatitis B core (HBc) antibody together with hepatitis B virus DNA (HBV-DNA)
  * Presence of hepatitis C ribonucleic acid (RNA)
* Known human immunodeficiency virus (HIV) infection. Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2026-05-18 (Estimated); Study Completion 2026-11-25 (Estimated)

PRIMARY OUTCOMES:
Mean relative change from baseline of [89Zr]Zr-BI 764532 tumour-to-plasma ratios in all detectable lesions post BI 764532 doses | at baseline and up to 35 days

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC Locatie VUMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com